CLINICAL TRIAL: NCT02625519
Title: Prospective, Randomized Open Trial to Evaluate the Efficacy of Highly Purified Urinary FSH Versus Recombinant FSH in Oocyte Donors Undergoing Controlled Ovarian Stimulation Based on Receptor N680S FSH Gene Polymorphism. Genodon Trial
Brief Title: Efficacy of Urinary Vs Recombinant FSH in Oocyte Donors Based on Receptor N680S FSH Gene Polymorphism (Genodon Trial)
Acronym: GENODON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Joaquín Llácer, Gynaecologist. Reproductive Medicine Specialist at Institute Bernabeu, Instituto Bernabeu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BER-FSH-2015-01; 2015-003779-31 (EudraCT Number)
Record Dates: First submitted 2015-11-09; First posted 2015-12-09 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Reproductive Techniques, Assisted
Keywords: Controlled ovarian stimulation; Follicle-stimulating hormone; Receptor N680S follicle-stimulating hormone receptor (FSHR); Gene polymorphism; Oocyte donors
MeSH Terms: conditions — Helping Behavior | interventions — Urofollitropin; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Urinary follicle-stimulating hormone (Experimental): Controled Ovarian stimulation with urinary follicle-stimulating hormone
  Interventions: Drug: Urinary follicle-stimulating hormone
- Recombinant follicle-stimulating hormone (Experimental): Ovarian stimulation with recombinant follicle-stimulating hormone
  Interventions: Drug: Recombinant follicle-stimulating hormone

INTERVENTIONS:
Drug: Urinary follicle-stimulating hormone — Ovarian stimulation with highly purified urinary follicle-stimulating hormone
  Other Names: urinary FSH; Fostipur®
  Arms: Urinary follicle-stimulating hormone
Drug: Recombinant follicle-stimulating hormone — Controled ovarian stimulation with recombinant follicle-stimulating hormone
  Other Names: recombinant FSH; Bemfola®
  Arms: Recombinant follicle-stimulating hormone

SUMMARY:
Exploratory, prospective, randomized, comparative, open trial with control group treated to assess whether the effective use of urinary FSH (uFSH) or recombinant FSH (rFSH) can be influenced by genotype of receptor N680S FSH Gene Polymorphism.

DETAILED DESCRIPTION:
The aim of this study is to determine whether the number of oocytes obtained in women oocyte donors may be different with the use of rFSH or uFSH based on receptor N680S FSHR gene polymorphism.

This is an exploratory, prospective, randomized, comparative, open trial with control group treated according to the usual therapeutic approach in our institution for ovarian stimulation for oocyte donors prospective exploratory study control group .

Three groups will be set based on follicle-stimulating hormone receptor (FSHR) genotype for the polymorphism N680: Group SS (Ser/Ser), group SN (Ser/Asn) and group NN (Asn/Asn). Donor members of each group will be randomly assigned to receive daily 225 IU of recombinant or urinary FSH for controlled ovarian stimulation protocol with antagonists. To avoid unintentional bias, allocation to treatment group will take place at the time in which ovarian stimulation according begins with a list of random allocation of treatments for each of the groups (SS , SN and NN) that will be associated the code of the patient and are prepared and will be available before the start of the study. The code assignment and treatment of the patient will consecutively in the order of the list and must be recorded in the medical history of the patient. The next scheduled patient will be assigned to the code and the next immediate treatment in this list.

The protocol for controlled ovarian stimulation in oocyte donors, will be performed always according to the usual protocol in the Instituto Bernabeu.

ELIGIBILITY:
Inclusion Criteria:

* Be considered eligible to get into the oocyte donation program of Instituto Bernabeu
* Age between 18 and 30 years
* Body Mass Index over 18 and under 28
* Antral follicle count greater than 9 and less than 25 (adding both ovaries)
* Patients starting ovarian stimulation with 225 IU of FSH
* Presence of both ovaries
* Ability to participate and comply with the study protocol
* Signing the written consent form
* Not having received treatment with ovulation stimulators in the 3 months prior to stimulation

Exclusion Criteria:

* Not suitable for inclusion in the oocyte donation program of Institute Bernabeu
* Concurrent participation in another study

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
number of cumulus-oocyte complexes obtained | through study completion, an average of 2 weeks
  number of cumulus-oocyte complexes obtained by follicle puncture at the end of ovarian stimulation

SECONDARY OUTCOMES:
number of metaphase II (MII) oocytes | through study completion, an average of 2 weeks
  number of metaphase II (MII) oocytes obtained by follicle puncture at the end of ovarian stimulation
number of useful oocytes (inseminated or microinjected) | through study completion, an average of 2 weeks
  number of useful oocytes after artificial insemination or microinjection
duration of stimulation (days) | through study completion, an average of 2 weeks
  mean number of days between the start of ovarian stimulation until the day of the follicular puncture
FSH treatment units obtained by oocyte | through study completion, an average of 2 weeks
  FSH treatment units administrated per oocyte obtained
FSH treatment cost per oocyte obtained | through study completion, an average of 2 weeks
  FSH treatment cost per oocyte obtained
fertilization rate | through study completion, an average of 2 weeks
  fertilization rate at 18 hours post-insemination
occurrence of side effects | through study completion, an average of 2 weeks
  occurrence of side effects associated with urinary FSH and recombinant FSH

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Llácer, Principal Investigator — Instituto Bernabeu
Locations (1):
- Instituto Bernabeu, Alicante, Spain